CLINICAL TRIAL: NCT04197804
Title: Do Mirror Neurons Play a Role in Tourette Syndrome Physiopathology? A Pilot Study.
Brief Title: Impulse Control in Gilles de la Tourette Syndrome
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: Nessie (PI: M Porta); L3035 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2018-12-29; First posted 2019-12-13 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tourette group: 20 subjects with Tourette Syndrome undergoing an evaluation to identify the IQ. Subsequently, 4 tasks are presented. The 1st (with a duration of about 2 and a half minutes) and the 2nd (with a duration of about 2 minutes) concerning the motor field, the 3rd (with duration of about 1 minute) and the 4th (with duration of about 3 minutes) concerning the linguistic field.
  Interventions: Other: Routine tests perform
- Control group: 20 subjects without Tourette Syndrome subjected to an evaluation to identify the IQ. Subsequently 4 tasks are presented. The 1st (with a duration of about 2 and a half minutes) and the 2nd (with a duration of about 2 minutes) concerning the motor field, the 3rd (with duration of about 1 minute) and the 4th (with duration of about 3 minutes) concerning the linguistic field.
  Interventions: Other: Routine tests perform

INTERVENTIONS:
Other: Routine tests perform — The subjects of the Tourette group and control group are subjected to routine tests performed at Tourette Center and Extrapyramidal Diseases. Both groups are initially subjected to an evaluation that aims to identify the IQ and therefore 4 tasks are presented. The 1st (with a duration of about 2 and a half minutes) and the 2nd (with a duration of about 2 minutes) related to the motor field, the 3rd (with duration of about 1 minute) and the 4th (with duration about 3 minutes) the language field. These evaluations are in practice at the Center for Tourette patients; the tasks will be administered to both groups.

SUMMARY:
The study intends to evaluate the role of Mirror Neurons in the determination of gestures, words, and repetitive vocalizations in subjects affected by Tourette's syndrome and to verify if these subjects are faster to assemble sounds, in phonology and morphology, than the non-pathological population.

ELIGIBILITY:
Inclusion Criteria:

TOURETTE GROUP

* Consecutive patients belonging to the Tourette Center
* Caucasian
* Italian mother-tongue
* Age between 6 and 10 years completed
* Male and female 4: 1 (16 males and 4 females)
* Diagnosis of Tourette's syndrome for at least 1 year
* Presence of a value of YGTSS> 50%

NOT GROUP TOURETTE

* Caucasian
* Italian mother-tongue
* Age between 6 and 10 years completed
* Male and female 4: 1 (16 males and 4 females)

Exclusion Criteria:

TOURETTE GROUP

* Diagnosis of DSA
* Presence of significant psychiatric disorders, with the exception of those belonging to the Tourette Syndrome itself (eg ADHD, OCD).

NOT GROUP TOURETTE

* Diagnosis of DSA
* Presence of significant psychiatric disorders

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The calculated sample size is 20 subjects per arm considering:
  1. error of I type with two queues = 0.05;
  2. Type II error β = 0.20, which corresponds to a test power (1-β = 0.80) of 80%;
  3. a clinically significant difference of 4%;
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Tourette syndrome and the imitation of gestures | Through study completion, an average of 1 year
  The aim is to investigate the correlation between Mirror Neurons and Tourette Syndrome defining the greater propensity of the Tourettian subjects to imitate gestures, through the administration of the first Task

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Porta, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy